CLINICAL TRIAL: NCT00750035
Title: Total Versus Subtotal Hysterectomy:a Randomised, Prospective Multicentre Study of the Effect on Urinary, Sexual and Bowel Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St George's Healthcare NHS Trust (Other)
Responsible Party: Ranee Thakar, St George's Healthcare NHS Trust
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 95.59.14
Record Dates: First submitted 2008-09-09; First posted 2008-09-10 (Estimated); Last update posted 2008-10-24 (Estimated); Status verified 2008-09

CONDITIONS: Hysterectomy
Keywords: Total hysterectomy; subtotal hysterectomy; urinary function; bowel function; sexual function; Quality of life; Psychological function

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): total abdominal hysterectomy and
  Interventions: Procedure: Total abdominal hysterectomy
- 2 (Experimental): Subtotal hysterectomy
  Interventions: Procedure: Subtotal abdominal hysterectomy

INTERVENTIONS:
Procedure: Total abdominal hysterectomy — Total abdominal hysterectomy and Subtotal abdominal hysterectomy
  Arms: 1
Procedure: Subtotal abdominal hysterectomy
  Arms: 2

SUMMARY:
Background

It is uncertain whether subtotal abdominal hysterectomy results in better bladder, bowel, or sexual function than total abdominal hysterectomy.

Methods

The investigators conducted a randomized, double-blind trial comparing total and subtotal abdominal hysterectomy in 279 women referred for hysterectomy because of benign disease; most of the women were premenopausal. The main outcomes were measures of bladder, bowel, and sexual function at 12 months. The investigators also evaluated postoperative complications.

ELIGIBILITY:
Inclusion Criteria:

* Women having abdominal hysterectomy for benign conditions of the uterus

Exclusion Criteria:

* Suspected cancer
* A body weight that exceeded 100 kg
* Previous pelvic surgery
* Known endometriosis
* Abnormal cervical smears,
* Symptomatic uterine prolapse
* Symptomatic urinary incontinence

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 279 (Actual)
Dates: Start 1996-01; Primary Completion 2000-04 (Actual); Study Completion 2000-04 (Actual)

PRIMARY OUTCOMES:
Main outcome measure was stress incontinence | Completed

SECONDARY OUTCOMES:
Quality of life | Completed

CONTACTS AND LOCATIONS:
Locations (1):
- St George's Healthcare NHS Trust, London, United Kingdom

REFERENCES:
- [Background] Thakar R, Ayers S, Clarkson P, Stanton S, Manyonda I. Outcomes after total versus subtotal abdominal hysterectomy. N Engl J Med. 2002 Oct 24;347(17):1318-25. doi: 10.1056/NEJMoa013336. PMID 12397189
- [Background] Thakar R, Ayers S, Georgakapolou A, Clarkson P, Stanton S, Manyonda I. Hysterectomy improves quality of life and decreases psychiatric symptoms: a prospective and randomised comparison of total versus subtotal hysterectomy. BJOG. 2004 Oct;111(10):1115-20. doi: 10.1111/j.1471-0528.2004.00242.x. PMID 15383114
- [Derived] Thakar R, Ayers S, Srivastava R, Manyonda I. Removing the cervix at hysterectomy: an unnecessary intervention? Obstet Gynecol. 2008 Dec;112(6):1262-1269. doi: 10.1097/AOG.0b013e31818f3bf5. PMID 19037034